CLINICAL TRIAL: NCT05839483
Title: A Single Center Study on the Evaluation of Diagnostic Efficacy of CXCR4 Targeted PET Imaging in Primary Aldosteronism
Brief Title: CXCR4 Targeted PET Imaging in APA Preoperative Localization Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Zhe Meng
Record Dates: First submitted 2023-03-24; First posted 2023-05-03 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-03

CONDITIONS: Aldosterone-Producing Adenoma
Keywords: Hypertension; Hypokalemia; Adrenal adenoma
MeSH Terms: conditions — Adrenocortical Adenoma; Hypertension; Hypokalemia; ACTH Syndrome, Ectopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4 (Experimental): scanned by 68Ga-PentixaFor PET imaging
  Interventions: Diagnostic Test: CXCR4

INTERVENTIONS:
Diagnostic Test: CXCR4 — Participants diagnosed with PA will be asked to be scanned by 68Ga-PentixaFor PET imaging.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of CXCR4 targeted PET imaging in preoperative localization diagnosis of primary aldosteronism (PA). Participants diagnosed with PA will be asked to be scanned by 68Ga-PentixaFor PET, and then underwent adrenal venous sampling (AVS). Then, the responsible adrenal adenoma will be resected by adrenalectomy, and examined with pathological section and staining. Researchers will compare the sensitivity and specificity between 68Ga-PentixaFor PET imaging and AVS in preoperative localization diagnosis of PA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PA, confirmed by an elevated aldosterone/renin ratio (ARR) and an intravenous salt loading test.
* The patient has provided written informed consent authorisation before participating in the study.
* The patient is 18 to 70 years of age at the time of consent.

Exclusion Criteria:

* Refusal by the patients to undergo 68Ga-PentixaFor PET/CT, AVS, CT, or adrenalectomy.
* Suspicion of familial hyperaldosteronism type 1 (FH-1) or type 3 (FH-3).
* Suspicion of adrenocortical carcinoma.
* Severe comorbidity potentially interfering with treatment or health-related quality of life.
* Patients need to take drugs that interfere with clinical research.
* Any medical condition present that in the opinion of the investigator will affect patients clinical status.
* Pregnancy or lactation.
* Estimated glomerular filtration rate <40mL/min/1.73m2.
* Interfering treatment in between 68Ga-PentixaFor PET/CT and AVS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
renin | immediately after admission
  measure the level of renin in blood
aldosterone | immediately after admission
  measure the level of aldosterone in blood
SUVmax | immediately after 68Ga-PentixaFor PET imaging
  measure the maximum standardized uptake value of adrenal adenoma, liver, and lateral normal adrenal
sensitivity | immediately after pathological examination
  the sensitivity of 68Ga-PentixaFor PET imaging in preoperative localization diagnosis of PA
specificity | immediately after pathological examination
  the specificity of 68Ga-PentixaFor PET imaging in preoperative localization diagnosis of PA
positive predictive value,PPV | immediately after pathological examination
  the PPV of 68Ga-PentixaFor PET imaging in preoperative localization diagnosis of PA
negative predictive value, NPV | immediately after pathological examination
  the NPV of 68Ga-PentixaFor PET imaging in preoperative localization diagnosis of PA

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Meng, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cui Y, Zhang Y, Ding J, Wang H, Ma X, Wang O, Chang X, Sun H, Huo L, Tong A. A Rare Aldosterone-Producing Adenoma Detected by 68Ga-pentixafor PET-CT: A Case Report and Literature Review. Front Endocrinol (Lausanne). 2019 Nov 29;10:810. doi: 10.3389/fendo.2019.00810. eCollection 2019. PMID 31849839
- [Result] Chaman Baz AH, van de Wiel E, Groenewoud H, Arntz M, Gotthardt M, Deinum J, Langenhuijsen J. CXCR4-directed [68Ga]Ga-PentixaFor PET/CT versus adrenal vein sampling performance: a study protocol for a randomised two-step controlled diagnoStic Trial Ultimately comparing hypertenSion outcome in primary aldosteronism (CASTUS). BMJ Open. 2022 Aug 23;12(8):e060779. doi: 10.1136/bmjopen-2022-060779. PMID 35998969
- [Result] Ding J, Zhang Y, Wen J, Zhang H, Wang H, Luo Y, Pan Q, Zhu W, Wang X, Yao S, Kreissl MC, Hacker M, Tong A, Huo L, Li X. Imaging CXCR4 expression in patients with suspected primary hyperaldosteronism. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2656-2665. doi: 10.1007/s00259-020-04722-0. Epub 2020 Mar 23. PMID 32206838